CLINICAL TRIAL: NCT07318038
Title: The Use of Rhythmic Light Therapy in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-25-01233
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dual frequency flickering light (Experimental): Light flickering with 10 Hz + 40 Hz visual stimulation
  Interventions: Device: Flickering Light
- Single frequency flickering light (Experimental): Light flickering with 10 Hz visual stimulation
  Interventions: Device: Flickering Light
- non-rhythmic flickering light (Placebo Comparator): Light flickering with random visual stimulation
  Interventions: Device: Flickering Light

INTERVENTIONS:
Device: Flickering Light — Red Flickering Light programed to three different visual stimulations

SUMMARY:
In this within-subjects, crossover study, participants will undergo Electroencephalogram (EEG) recordings before, during, and after each of three 1-hour sessions. All participants will experience all three conditions: (1) dual-frequency visual (10 and 40 Hz), (2) single-frequency visual (40 Hz), and (3) non-rhythmic stimulation. EEG spectral power and amplitude coupling will be analyzed to determine whether stimulation-induced increases in alpha-gamma neural synchrony translate to improvements in cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* History of Mild Cognitive Impairment with a Montreal Cognitive Assessment score between 18 and 25

Exclusion Criteria:

* History of epilepsy or photosensitivity
* Blindness or other obstructive vision conditions
* retinal diseases
* presence of another brain disease accounting for their cognitive status

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
EEG-based neural synchrony | 5 minute EEG recording will be done at start, middle and end of each one-hour session, each session separated by one week
  Change in spectral power and amplitude in the alpha and gamma EEG bands. Increase in power and amplitude is indicative of increases in neural synchrony.

SECONDARY OUTCOMES:
Digit Span Task | Completed at start and end of each one-hour session, each session will be separated by one week
  Change in cognition will be measured by the Digit Span Task which is a working memory task. Increase in accuracy and response time indicates improved cognitive performance.
  Digit Span. Memory span is the longest list of items that a person can repeat back in correct order immediately after presentation on 50% of all trials. Items may include words, numbers, or letters. The task is known as digit span when numbers are used. Memory span is a common measure of short-term memory. A digit-span task is used to measure working memory's number storage capacity. The item score is the sum of the scores on the two trials for that item (range=0-2). The total raw score for backwards digit span is the sum of the item scores; maximum backwards digit span total raw score is 16 points. Higher score indicates better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
As the primary outcome measure of this study is EEG recordings, individual results will not be shared.